CLINICAL TRIAL: NCT04189328
Title: Clinical and Radiological Comparison of Peri Implant Soft Tissue Parameters and Crestal Bone Loss Around Microsurgically and Macrosurgically Placed Implants: A Randomised Controlled Clinical Trail
Brief Title: Peri-implant Papillary Height Comparison in Microsurgically and Macrosurgically Placed Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_82168
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Dental Implants

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): conventional macrosurgical implant placement
  Interventions: Procedure: macrosurgical dental implant placement
- test group (Experimental): microsurgical implant placement
  Interventions: Procedure: dental implant placement using magnifying loupes and microsurgical instruments

INTERVENTIONS:
Procedure: dental implant placement using magnifying loupes and microsurgical instruments — microsurgical dental implant placement employin splt finger technique by Misch
  Arms: test group
Procedure: macrosurgical dental implant placement — macrosurgical placement of single dental implants
  Arms: control group

SUMMARY:
This study compares the peri-implant soft tissue and crestal bone loss around single implants when placed macrosurgically and microsurgically.

DETAILED DESCRIPTION:
Black triangles in dentition especially in the anterior teeth would pose an esthetic concern. Interdental papilla height is crucial for eliminating this black triangle.

32 participants, 16 in two groups were assigned randomly. Microsurgical approach using microsurgical instruments and magnifying loupes were used for one group participants and similar procedure without magnifying loupes and microsurgical instruments was done in the other group.

comparsion of the microsurgical outcome is done by measuring peri implant papilla gain and radiographic crestal bone loss will be done between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients desiring implant placement for replacement of missing tooth and willing to participate in the study

  * Non smokers
  * Patients who do not report any relevant medically comprimising conditions or had not received any radiation therapy in head and neck region for cancer therapy.
  * Subjects with satisfactory residual ridges who demonstrated adequate bucco-lingual and mesio-distal space for implant placement, that facilitates primary stability.
  * Patients who demonstrate Plaque Index <10% and good compliance.
  * Full mouth bleeding scores ≤25% before the implant placement.
  * Sites with sufficient band of keratinised mucosa.

Exclusion Criteria:

* • Pregnant and lactating females

  * Patients on anticancer therapy and immunosuppressant drugs.
  * Implants to be placed in sites with previous periodontal disease
  * Bleeding disorder or on anticoagulant therapy
  * Systemic diseases that would negatively influence wound healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
peri-implant papilla height | 1 year
  mesial and distal peri implant papilla height is measured in millimeter
marginal gingiva | 1 year
  buccal marginal gingival height is measured
jemt papilla index | 1 year
  papillary height gained around implant is scored using jemt papilla index 0 = no papilla and no indication of a curvature of the soft tissue adjacent to the implant crown are present;
  1. = less than one-half of the papilla height is present, and a convex curvature of the soft tissue adjacent to the implant crown and adjacent tooth can be observed;
  2. = at least one-half of the papilla height is present but not to the contact point between the teeth, the papilla is not completely harmonious with the adjacent papillae between the permanent teeth, and soft tissue is harmonious with adjacent teeth;
  3. = the papilla fills the entire proximal space and is harmonious with the adjacent papillae, and soft-tissue contour is optimal;
  4. = the papillae are hyperplastic and cover too much of the implant or the adjacent tooth, and the soft-tissue contour is irregular
crestal bone loss | 1 year
  radiographic crestal bone level around the implants measured from 1st thread of the implant to the coronal or apical most bone level in millimeters.
pink esthetic score | 1 year
  scoring assigned to 7 soft tissue criteria by an examiner as 0,1,2,3 and the average of the total score is considered the final score. a maximum score of 14 can be alloted

SECONDARY OUTCOMES:
surgical time taken | 1 day
  the time taken right from the incision to the implant placement is watched and recorded.
visual analogue scale score | 1 year
  aesthetic score by the outcome investigator using VAS score sheet of 10 points. 1 being most painful and 10 being painless
probing depth | 1 year
  peri implant probing depth at each follow up was recorded
plaque index | 1 year
  plaque scores were recorded at each follow up 0.-0.9 good 1.0-1.9-fair 2-3-poor
gingival index | 1 year
  gingival index scores were recorded at each followup 0.1-1-mild gingivitis 1.1-2- moderate gingivitis 2.1-3 severe gingivitis

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Joann pauline George, MDS, Principal Investigator — Krishnadevaraya college of dental sciences
Locations (1):
- Krishnadevaraya college of dental sciences and hospital, Bangalore, Karnataka, India